CLINICAL TRIAL: NCT03434938
Title: Motivational Intervention for Older Adults Undergoing Inpatient Post-stroke Geriatric Rehabilitation and in Transition to Home
Brief Title: IMAGINE Study Protocol
Acronym: IMAGINE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Parc Sanitari Pere Virgili (Other)
Collaborators: Vall d'Hebron Institute of Research (Unknown); Health and Ageing Foundation of the Autonomous University of Barcelona (Unknown); Center for Ageing and Supportive Environments (Unknown); Hospital Universitari de Santa Maria (Unknown); Consorci Sanitari Integral (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IMAGINE (ID 373 / 49)
Record Dates: First submitted 2018-01-23; First posted 2018-02-15 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Patients (>=60 Years Old) Suffering From Mild-moderate Stroke (Ischemic or Hemorrhagic, Stroke Severity Assessed by NIHSS <16 Points)
Keywords: Stroke; Geriatric; Rehabilitation; Functional recovery; Physical activity; Motivational interviewing; Adherence; Clinical trial
MeSH Terms: conditions — Ischemia; Stroke; Motor Activity | interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: MI intervention will be associated to standard geriatric rehabilitation. MI will be structured in 4 sessions (within 72 hours from admission, within next 6 days after first MI session, at 1 week from the second session and pre-discharge), with the goals of reducing disability obtaining patients' collaboration, creating a shared tailored plan which would complement the individual approach established by the multidisciplinary team as part of routine geriatric rehabilitation unit, and reinforcing engagement and adherence at 3 months.
  Standard rehabilitation and control includes a multidisciplinary and individualized treatment plan based on comprehensive geriatric and specific rehabilitation assessments.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: After inclusion in the study and obtaining informed consent, participants will be randomized to intervention or control group in a concealed allocation manner. Centralized randomization will be conducted through a block randomization procedure, with random-varying block size, stratified by participating centre. Participants will be randomized after the baseline assessment, guaranteeing the blinded assessment. The 30 days and 3 months assessments will be conducted by an assessor blinded to participants' group allocation, who will ask the participants not to disclose their group allocation. Afterwards, the assessor will record whether he/she was made aware of the participant allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MI Intervention (Experimental): Standard geriatric rehabilitation combined with 4 MI sessions (within 72 hours from admission, within 6 days, at 1 week from the second session and pre-discharge, respectively). MI will be delivered by nurses trained through a certified MI course and additional group coaching sessions will be offered them throughout the study. Quality control of the MI sessions will be carried out using Motivational Interviewing Treatment Integrity (MITI) Code 3.1.1 through random video recording.
  Interventions: Behavioral: Motivational interviewing
- Standard rehabilitation (No Intervention): Routine geriatric rehabilitation will include a multidisciplinary and individualized treatment plan based on comprehensive geriatric and specific rehabilitation assessments. As a specific control intervention, within 72 hours from admission a nurse without training in MI will handle the patient written information about generic benefits of exercising.

INTERVENTIONS:
Behavioral: Motivational interviewing — MI sessions' goals will to obtain patients' collaboration, creating a shared tailored approach to complement the individual geriatric rehabilitation plan, and reinforcing engagement and adherence at 3 months.
  All 20-minutes sessions will follow the logical sequence of MI by Rollnick and Millner (engaging, focusing, evoking and planning) in a semi-structured format to ensure homogeneity. Content will include: 1) Creating engagement with patients by exploring their preferences, values, goals, and their knowledge and expectations about rehabilitation and recovery, 2) enhancing motivation by evoking patients' strengths and abilities, 3) follow-up and reinforcement, and 4) adapting the plan to the improved abilities and to home setting after discharge.
  Arms: MI Intervention

SUMMARY:
Background: Rehabilitation pathways are crucial to reduce stroke-related disability. Motivational Interviewing (MI), a centred-person intervention aimed to empower and motivate the patient, could be a resource to improve rehabilitation and its outcomes for older stroke survivors.

Objective: The IMAGINE project aims to assess the impact of MI associated to standard geriatric rehabilitation, on 30 days functional improvement measured by the Functional Independence Measure (FIM), compared to standard geriatric rehabilitation alone, in patients admitted to geriatric rehabilitation after a stroke. Secondary objectives will be to assess the impact on physical activity and performance, self-efficacy, sense of coherence, safety, cost-utility and participants' experience, plus functional status at 3 months.

Methods: Multicenter randomized clinical trial in three geriatric rehabilitation departments. Older adults after mild-moderate stroke without previous dementia, post-stroke severe cognitive impairment or delirium at admission, severe previous disability, aphasia or terminal conditions will be randomized into the control or the intervention group (136 per group, total N = 272). The control group will receive written information about the benefits of exercising, besides standard rehabilitation. The intervention group, in addition, will receive 4 sessions of MI by trained nurses. A shared tailored plan based on patients' goals, needs, preferences and capabilities will be agreed. Besides the FIM, in-hospital physical activity will be measured through accelerometers (activPAL) and secondary outcomes using internationally validated scales. As a complex intervention, a process evaluation and cost-utility assessments will be performed too.

Results: Final results are expected by end of 2020. Implications: This project aims to achieve impacts on functional status, disability and physical performance and behavioral (increasing physical activity) and psychological implications (on general self-efficacy and sense of coherence) through a non-pharmacological and likely accessible, acceptable and scalable intervention. Efficiency and value, based on costs/quality adjusted life years, will be assessed. Moreover, a reduction in post-stroke disability would have social benefits also for families and would reduce health and social care costs. In brief, advances will be in terms of a better rehabilitation process.

DETAILED DESCRIPTION:
IMAGINE project aims to investigate the effect of adding an adapted MI approach to the usual geriatric rehabilitation to motivate and empower stroke patients to participate in their own rehabilitation plan and thus, to increase their physical activity and engagement in self-care and other activities. The main aim is to finally improve patients' physical and global function and, in turn, to reduce dependency. As mentioned, there is evidence-base around MI in rehabilitation, which covers functional, clinical and efficiency aspects. It is expected that IMAGINE project will add a relevant contribution for the implementation of this intervention in older adults with post-stroke residual disability and dependency needing rehabilitation. Accordingly, this study should inform practice and policy on how to move forward towards shared decision making and shared responsibilities in a vulnerable population such as older adults with a recent stroke.

ELIGIBILITY:
Inclusion criteria:

1. Older adults (>=60 years old).
2. Admitted to the geriatric rehabilitation hospital after a mild-moderate stroke (ischemic or hemorrhagic); stroke severity assessed by National Institute of Health Stroke Severity (NIHSS) scale <16 points.
3. Able to provide informed consent.

Exclusion Criteria:

1. Previous diagnosis of dementia (ascertained from medical records).
2. Moderate-severe post-stroke cognitive impairment (Pfeiffer SMPQ>7 errors) or persistent delirium after 7 days from admission.
3. Previous severe disability in the activities of daily living (pre-stroke Barthel index <20/100 points).
4. Severe stroke which might limit recovery (NIHSS>=16).
5. Aphasia or other problems which limit communication and 6) advanced and terminal condition (prognosis not exceeding 6 months).

Ages: 60 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Estimated)
Dates: Start 2018-06-19 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Functional Independence Measure (FIM). | At admission (within 72 hours), 30 days, and at 3 months follow-up.
  The FIM is used to track functional evolution during in-hospital rehabilitation process. FIM is comprised of 18 items, grouped into 2 subscales: 1) motor and 2) cognition. The motor subscale includes: Eating, grooming, bathing, dressing (upper body), dressing (lower body), toileting, bladder management, bowel management, transfers (bed/chair/wheelchair), transfers (toilet), transfers (bath/shower), walk/wheelchair, stairs. The cognition subscale includes: Comprehension, expression, social interaction, problem solving, memory. The total score for the FIM instrument (the sum of the motor and cognition subscale scores) will be a value between 18 and 126. The higher the score, the more independent the patient is in performing the task associated with that item.

SECONDARY OUTCOMES:
Modified-Rankin Scale (mRS) | At admission (within 72 hours; recall period, previous to event), and at 3 months follow-up.
  The Modified Rankin Scale (mRS) assesses disability in post-stroke patients and it can be used to track functional evolution over time. A score of 0 is "no disability", 5 is "disability requiring constant care for all needs" and 6 is "death".
The Canadian Performance Oriented Measure (COPM). | At 30 days from admission, and at 3 months follow-up.
  The COPM is a semi-structure interview that enables patient to identify problems and priorities in the three areas of occupational performance: self-care, productivity, and leisure. Once problems have been identify, patient needs to rate them using a 10-point scale. Then, patient will need to pick up to 5 most important problems to work. Finally, two subscale scores are obtained: performance (COPM-P) and satisfaction with performance (COPM-S).
In-hospital physical activity. | 7 consecutive in-hospital days after admission, preferably within 10 days before discharge.
  This will be measured through accelerometers (ActivPAL) located at the preserved leg, to measure mainly time spent sitting and standing.
Short Physical Performance Battery (SPPB). | At admission (within 72 hours), 30 days, and at 3 months follow-up.
  Improvement in physical performance will be measured using the SPPB, including balance, strength and gait velocity sub-items.
Number of adverse events registration. | At 30 days after admission, and at 3 months follow-up.
  The incidence of diverse adverse events will be registered (yes vs. no; and number of times occuring each incident). Variables collected are: Falls, fractures, cranial traumatism, cardiovascular events (specifically: angina, myocardial infarction, TIA, stroke), aspiration pneumonia/respiratory infections, readmissions to acute hospitals and death. A final composite (total number of adverse events for each patient) will be obtained.
Self-perceived pain: 10-point numeric scale | At 30 days after admission, and at 3 months follow-up.
  Self-perceived pain will be assessed by means of a 10-point numeric scale (0 = no pain at all, 10 = worst possible pain).
General Self-Efficacy scale (GSE). | At 30 days after admission, and at 3 months follow-up.
  The GSE is a 10-item tool designed to assess optimistic self-beliefs to cope with a variety of difficult demands in life. This scale is correlated to emotion, optimism and work satisfaction. Negative coefficients are found for depression, stress, health complaints, burnout, and anxiety. The total score is calculated by finding the sum of the all items. For the GSE, the total score ranges between 10 and 40, with a higher score indicating more self-efficacy.
Sense of coherence (SOC) questionnaire. | At 30 days after admission, and at 3 months follow-up.
  SOC-13 has three components: Comprehensibility, Manageability and Meaningfulness. This scale is rated on a 7-point likert scale, a total score can also be used. The mean alpha of the SOC-13 scale was .82 (range = .74 - .81).
Process variables - Length of hospital stay. | Through study completion, an average of 40 days.
  Length of stay (total numer of days) for each patient will be measured considering as an endpoint patients' hospital discharge.
Process variables - Destination at discharge. | Through study completion, an average of 40 days.
  Discharge destination (specifically: home, nursing home, long-term care, acute hospital, death) will be registered for each patient.
Process variables - Total time of rehabilitation. | Through study completion, an average of 40 days.
  Total time of rehabilitation (total numer of days) will be registered for each patient.
Cost-utility measures. | At admission (within 72 hours), 30 days, and at 3 months follow-up.
  Cost-utility will be measured as the ratio between direct costs during hospitalization (considering costs that include workforce time use, exams, use of other hospital resources, visits) and Quality Adjusted Life Years (QALYs) obtained by means of the EQoL-5D administered before and after the treatment.
  Cost-utility will be calculated as the incremental ratio €/QALYs in the intervention vs. control group.
Rehabilitation efficiency. | Through study completion, an average of 40 days.
  Rehabilitation efficiency scores for each patient will be computed as the improvement in the FIM/length of hospital stay.

OTHER OUTCOMES:
Participants perceptions and experiences of the intervention. | At 30 days of hospitalization, and at 3 months follow-up.
  Qualitative evaluation will be aimed to explore participant's experiences in the frame of the process evaluation of the intervention. Process evaluation will be based on MRC guidance, and will focus on how the context, implementation and impact mechanisms will influence the results. In particular, participants' experiences, their perceived impacts as well as unexpected effects will be explored through in-depth interviews at 30 days and at 3 months on a purposeful sample of participants, selected to maximize variability (by gender, disability levels, socio-economic levels, and social support). In addition, a purposeful sample of caregivers and professionals who performed the intervention will be also interviewed and we will conduct a focus group with reference professionals of the wards.

CONTACTS AND LOCATIONS:
Locations (6):
- Spain (5):
  - Fundació Salut i Envelliment Universitat Autònoma de Barcelona, Bellaterra, Barcelona
  - Consorci Sanitari Integral - Hospital General de L'Hospitalet & Hospital de St Joan Despí, L'Hospitalet de Llobregat, Barcelona
  - Parc Sanitari Pere Virgili, Barcelona
  - Hospital Universitari Vall d'Hebron - Fundació Institut de Recerca Vall d'Hebron, Barcelona
  - Hospital Universitari Santa Maria, Lleida
- University of Lund, Lund, Sweden

REFERENCES:
- [Derived] Gual N, Perez LM, Castellano-Tejedor C, Lusilla-Palacios P, Castro J, Soto-Bagaria L, Coll-Planas L, Roque M, Vena AB, Fontecha B, Santiago JM, Lexell EM, Chiatti C, Iwarsson S, Inzitari M. IMAGINE study protocol of a clinical trial: a multi-center, investigator-blinded, randomized, 36-month, parallel-group to compare the effectiveness of motivational interview in rehabilitation of older stroke survivors. BMC Geriatr. 2020 Sep 4;20(1):321. doi: 10.1186/s12877-020-01694-6. PMID 32887564